CLINICAL TRIAL: NCT01822587
Title: Enhancing Disrupted Reconsolidation: Impact on Cocaine Craving, Reactivity and Use
Brief Title: Enhancing Disrupted Reconsolidation: Impact on Cocaine Craving
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21392
Record Dates: First submitted 2013-03-19; First posted 2013-04-02 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Cocaine Addiction
Keywords: Drug Abuse; Cocaine; Addiction
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Behavior, Addictive | interventions — Propranolol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Administered once orally following cue exposure on each of the first two days of testing.
  Interventions: Drug: Placebo
- Propranolol 40mg (Active Comparator): Administered once orally following cue exposure on each of the first two days of testing.
  Interventions: Drug: Propranolol, 40 mg
- Propranolol, 80mg (Active Comparator): Administered once orally following cue exposure on each of the first two days of testing.
  Interventions: Drug: Propranolol, 80 mg

INTERVENTIONS:
Drug: Propranolol, 40 mg
  Other Names: Inderal
  Arms: Propranolol 40mg
Drug: Propranolol, 80 mg
  Other Names: Inderal
  Arms: Propranolol, 80mg
Drug: Placebo
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The investigators' recently completed study has provided the first evidence that administration of the medication propranolol, following exposure to cocaine cues, can alter drug-associated memories and reduce craving and other drug cue-elicited responses in cocaine addicted persons. The investigators will attempt to augment this effect by a) doubling the number of propranolol-medicated cocaine cue exposure (CCE) retrieval sessions and b) increasing the dose of propranolol. It is expected that propranolol treated groups, relative to placebo treated groups, will evidence greater reduction of craving, cue reactivity and cocaine use during follow-up cocaine cue exposures. Also, these effects will be greater for those who receive 80mg of propranolol as opposed to 40mg.

DETAILED DESCRIPTION:
Three groups of CD (cocaine dependant) participants will receive two sessions of cocaine cue exposure (CCE), each separated by a 24 hr. period and both conducted while the participants remain in hospital. One group (PBO) will receive placebo following each CCE session while the second (40PP) and third (80PP) group will receive 40 mg and 80 mg propranolol, respectively. Participants will return two days, and 1, 3, and 6 weeks after discharge and will be administered a CCE session to assess for maintenance/generalization of disruption of reconsolidation (DoR) effects on craving and cue reactivity to familiar and novel cocaine cues. Participants will also be assessed 3 times weekly for cocaine use (self-report & urine drug screen) during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet DSM-IV criteria for current cocaine dependence (within the past month). Participants may meet criteria for abuse, but not dependence, for any other substance with the exception of nicotine. Because of the high comorbidity of cocaine and nicotine dependence, excluding nicotine dependence would seriously compromise the feasibility of recruitment (nicotine patch will be provided to participants during the course of their involvement in the laboratory procedures). Although individuals who meet criteria for alcohol abuse will be accepted for study participation, anyone who has a measurable blood alcohol level on the day of testing will be excluded as acute alcohol intake can lower seizure threshold.
* Participants must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.Exclusion Criteria:
* Use of one of the following methods of birth control by female participants: barrier methods (diaphragm or condoms with spermicidal or both), surgical sterilization, use of an intra-uterine contraceptive device, or complete abstinence from sexual intercourse.
* Individuals must live within a 50-mile radius of our research program and have reliable transportation.
* Individuals must consent to remain abstinent from all drugs of abuse (except nicotine) for 72 hours immediately prior to CTRC inpatient admission.
* Individuals must consent to random assignment to one of three study groups (the two propranolol-treated groups or the placebo-treated group).

Exclusion Criteria:

* Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
* Individuals with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect heart rate or skin conductance measurement.
* Individuals with significant liver impairment as propranolol is hepatically metabolized.
* Individuals with a history of or current psychotic disorder, current major depressive disorder, bipolar affective disorder or a severe anxiety disorder as these may impact cue reactivity.
* Individuals currently taking anti-arrythmic agents, psychostimulants or any other agents known to interfere with heart rate and skin conductance monitoring.
* Known or suspected hypersensitivity to propranolol.
* Individuals taking medications that could adversely interact with the study medication, including, but not limited to albuterol, insulin, or significant inhibitors of CYP2D6.
* Individuals with bronchial asthma or chronic obstructive pulmonary disease, as the use of propranolol is contraindicated in these individuals.
* Individuals with any physical condition or disability that would compromise optimal sensory processing of the cues (e.g., blindness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Saladin, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Administered once orally following cue exposure on each of the first two days of testing.
  Placebo
- Propranolol 40mg: Administered once orally following cue exposure on each of the first two days of testing.
  Propranolol, 40 mg
- Propranolol, 80mg: Administered once orally following cue exposure on each of the first two days of testing.
  Propranolol, 80 mg
Period: Overall Study
Arm/Group | Placebo | Propranolol 40mg | Propranolol, 80mg
Started (Not all participant who were started were able to complete the study.) | 59 | 60 | 62
Completed | 43 | 45 | 44
Not Completed | 16 | 15 | 18
Not completed — Lost to Follow-up | 7 | 9 | 12
Not completed — Physician Decision | 9 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Propranolol 40mg | Propranolol, 80mg | Total
Number analyzed (Participants) | 59 | 60 | 62 | 181
Age, Continuous [Mean (Full Range); unit: years] | 44.8 [21 to 69] | 43.8 [21 to 65] | 42.3 [19 to 59] | 43.6 [19 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 25 | 64
  Male | 39 | 41 | 37 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 22 | 19 | 19 | 60
  African American | 34 | 40 | 42 | 116
  Mixed/Unknown | 3 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 59 | 60 | 62 | 181

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use
Description: Timeline of cocaine use throughout the duration of the study (in dollar amounts)
Time Frame: Evaluated at Weeks 1, 3 and 6
Measure: Mean (Standard Error); unit: Dollar amounts of cocaine use
Arm/Group | Placebo | Propranolol 40mg | Propranolol, 80mg
Number analyzed (Participants) | 59 | 60 | 62
Dollar amounts of cocaine use
  Week 1 | 58.9 (31.95) | 71.57 (31.63) | 69.63 (30.74)
  Week 3 | 121.25 (32.67) | 177.67 (32.34) | 135.81 (31.93)
  Week 6 | 186.57 (33.21) | 198.9 (32.85) | 242.79 (32.47)

2. Primary Outcome: Change in Craving Score
Description: The participant is asked, "What is the level of craving you are experiencing on a scale or 0 to 100, with 0 representing no craving and 100 extreme craving"?
Time Frame: Single-Item Craving Scores are collected at all Retrieval Extinction Sessions (medication days), as well as all Phase Two Test Sessions (weeks 1,3 and 6).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Propranolol 40mg | Propranolol, 80mg
Number analyzed (Participants) | 59 | 60 | 62
score on a scale
  Day 2 | 25.6 (3.0) | 31.4 (2.9) | 26.9 (2.9)
  Week 1 | 27.5 (2.8) | 28.0 (2.8) | 24.7 (2.7)
  Week 3 | 24.6 (2.9) | 29.0 (2.9) | 20.0 (2.9)
  Week 6 | 22.6 (2.8) | 22.4 (2.7) | 17.5 (2.8)

3. Primary Outcome: Days of Abstinence
Description: How many days the participants used cocaine versus how many days of abstinence they were able to achieve.
Time Frame: Week 1, Week 3, and Week 6
Measure: Number; unit: Days
Arm/Group | Placebo | Propranolol 40mg | Propranolol, 80mg
Number analyzed (Participants) | 59 | 60 | 62
Days
  Week 1 | 20 | 19 | 17
  Week 3 | 15 | 14 | 13
  Week 6 | 15 | 9 | 7

4. Primary Outcome: Average Peak Craving Score
Description: Peak Craving Response from Session Baseline- peak craving is measured by a scale with a score of 0 (no craving) -100 (maximum craving).
Time Frame: Day 2, Week 1, Week 3, and Week 6
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Propranolol 40mg | Propranolol, 80mg
Number analyzed (Participants) | 59 | 60 | 62
score on a scale
  Day 2 | 16.1 (3.5) | 23.3 (3.4) | 18.1 (3.3)
  Week 1 | 15.2 (3.5) | 19.6 (3.5) | 17.1 (3.5)
  Week 3 | 13.1 (3.6) | 19.7 (3.6) | 10.1 (3.5)
  Week 6 | 10.2 (3.6) | 12.1 (3.6) | 5.5 (3.7)

5. Primary Outcome: Use Days
Description: Mean Days of Cocaine Use
Time Frame: Week 1, Week 3, Week 6
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | Propranolol 40mg | Propranolol, 80mg
Number analyzed (Participants) | 59 | 60 | 62
Days
  Week 1 | 1.66 (0.54) | 1.61 (0.53) | 1.76 (0.52)
  Week 3 | 3.33 (0.55) | 3.15 (0.54) | 3.51 (0.54)
  Week 6 | 4.9 (0.56) | 4.49 (0.55) | 6.06 (0.55)

ADVERSE EVENTS:
Time Frame: Adverse events will be monitored throughout the study (six weeks) and all events will be followed to resolution or stabilization.
Description: A serious adverse event is one that meets any of the following criteria:
  1. Fatal or life threatening
  2. Requires or prolongs inpatient hospitalization
  3. Results in persistent or significant disability/incapacity
  4. Congenital anomaly
  5. Medical event that may jeopardize the participant or require intervention to mitigate serious outcome
  6. Cancer
  7. Overdose
Arm/Group | Placebo | Propranolol 40mg | Propranolol, 80mg
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/60 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60 | 0/62
Other Adverse Events (participants affected / at risk) | 0/59 | 1/60 | 0/62
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=59) | Propranolol 40mg (N=60) | Propranolol, 80mg (N=62)
Participant Hospitalization (Psychiatric disorders) | 0 (0) | 1/1 (1) | 0 (0) — Participant was hospitalized for depression and suicidal thoughts (no attempt).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT01822587/Prot_SAP_000.pdf